CLINICAL TRIAL: NCT00184275
Title: Brain Metastases Tissue Characterized by High-resolution Magic Angle Spinning MR and Micro Array
Brief Title: Characterization of Brain Metastases
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12621
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Neoplasm Metastasis; Lung Neoplasms; Breast Neoplasms; Melanoma
Keywords: Brain metastasis; HR MAS spectroscopy; Tissue micro array; DNA micro array
MeSH Terms: conditions — Neoplasm Metastasis; Lung Neoplasms; Breast Neoplasms; Melanoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen tumor tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose is to characterize tumour biological markers in brain metastases tissue from patients with different primary tumour by using ex vivo techniques as high-resolution magic angle spinning MR spectroscopy and micro array.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of brain metastases

Exclusion Criteria:

* children
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with brain metastases
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Lundgren, MD PhD, Study Director — Cancer Clinic, St.Olavs Hospital Trondheim University Hospital; Ingrid S Gribbestad, PhD, Study Chair — Norwegian University of Science and Technology, Faculty of Medicine
Locations (1):
- Norwegian University of Science and Technology, Faculty of Medicine, Trondheim, Norway

REFERENCES:
- [Background] Sjobakk TE, Johansen R, Bathen TF, Sonnewald U, Kvistad KA, Lundgren S, Gribbestad IS. Metabolic profiling of human brain metastases using in vivo proton MR spectroscopy at 3T. BMC Cancer. 2007 Jul 27;7:141. doi: 10.1186/1471-2407-7-141. PMID 17662122
- [Result] Sjobakk TE, Vettukattil R, Gulati M, Gulati S, Lundgren S, Gribbestad IS, Torp SH, Bathen TF. Metabolic profiles of brain metastases. Int J Mol Sci. 2013 Jan 22;14(1):2104-18. doi: 10.3390/ijms14012104. PMID 23340650